CLINICAL TRIAL: NCT05495061
Title: A Phase III, Randomized, Observer-Masked, Active-Controlled, Parallel-Group, Multicenter Study Assessing the Efficacy and Safety of STN1012600 Ophthalmic Solution 0.002% Compared With Latanoprost 0.005% in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension (Angel-J1 Study)
Brief Title: A Comparative Confirmatory Study of STN1012600 in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101260005LT
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Primary Open Angle Glaucoma, Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STN1012600 0.002% (Experimental)
  Interventions: Drug: STN1012600 ophthalmic solution 0.002%
- Latanoprost 0.005% (Active Comparator)
  Interventions: Drug: Latanoprost ophthalmic solution 0.005%

INTERVENTIONS:
Drug: STN1012600 ophthalmic solution 0.002% — 1 drop STN1012600 ophthalmic solution 0.002% once daily for 3 months
  Arms: STN1012600 0.002%
Drug: Latanoprost ophthalmic solution 0.005% — 1 drop Latanoprost ophthalmic solution 0.005% once daily for 3 months
  Arms: Latanoprost 0.005%

SUMMARY:
To investigate whether the IOP lowering efficacy of STN1012600 ophthalmic solution 0.002% is non-inferior to that of latanoprost 0.005% in subjects with POAG or OHT after treatment for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Diagnosis of POAG or OHT in both eyes, or one eye with POAG and the other with OHT.
* Corrected Visual Acuity of +0.60 logMAR (Decimal visual acuity 0.3) or better in each eye.

Exclusion Criteria:

* Presence of any active severe external ocular disease, inflammation, or infection of the eye and/or eyelids in either eye.
* History of severe ocular trauma in either eye.
* Any condition that prevents clear visualization of the fundus in either eye.
* Known allergy, hypersensitivity or contraindications to any components of the study medications or other study related procedures/medications.
* History of ocular surgery specifically intended to lower IOP in either eye.
* History of keratorefractive surgery in either eye.
* Females who are pregnant, nursing, or planning a pregnancy.
* Subjects with known or suspected drug or alcohol abuse.
* Participation in other investigational drugs or device clinical trials within 30 days prior to Screening.
* Any decision by the Investigator to terminate a subject in screening or declare any subject ineligible for any sound medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean diurnal intraocular pressure | 4 weeks
  Change from baseline in mean diurnal intraocular pressure at Week 4

CONTACTS AND LOCATIONS:
Locations (44):
- Japan (44):
  - Eyecare Nagoya, Aichi
  - Kitanagoya Eye Clinic, Aichi
  - Takahashi Eye Clinic, Aichi
  - Kawabata Eye Clinic, Chiba
  - Mitsuhashi Eye Clinic, Chiba
  - Shisui Ophthalmology Clinic, Chiba
  - Takeda Eye Clinic, Hokkaido
  - Kanamori Eye Clinic, Hyōgo
  - Dannoue Eye Clinic, Kanagawa
  - Hodogaya iina Eye Clinic, Kanagawa
  - Honda Eye Clinic, Kanagawa
  - Yokosuka Chuoh Eye Clinic, Kanagawa
  - Kengun Sakuragi Eye Clinic, Kumamoto
  - Hideyuki Eye Clinic, Miyagi
  - Iwashita Eye Clinic, Osaka
  - Maeda Eye Clinic, Osaka
  - Nishi Eye Hospital, Osaka
  - OCROM Clinic, Osaka
  - Onoe Eye Clinic, Osaka
  - Sugasawa Eye Clinic, Osaka
  - Sugiura Eye Clinic, Osaka
  - Tahara Eye Clinic, Osaka
  - Tane Memorial Eye Hospital, Osaka
  - Kawaguchi Aozora Eye Clinic, Saitama
  - Omiya Hamada Eye Clinic West entrance Branch, Saitama
  - Omiya Hamada Eye Clinic, Saitama
  - Shibuya Ophthalmology Clinic, Saitama
  - Muramatsu Eye Clinic, Shizuoka
  - Nakamura Eye Clinic, Shizuoka
  - Ono Ophthalmic Clinic, Shizuoka
  - Saito Eye Clinic, Shizuoka
  - Yoshimura Eye & Internal Medical Clinic, Shizuoka
  - Dogenzaka Kato Eye Clinic, Tokyo
  - Hashida Eye Clinic, Tokyo
  - Kakinoki Eye Clinic, Tokyo
  - Seijo Clinic, Tokyo
  - Shimizu Eye Clinic, Tokyo
  - Shirayama Eye Clinic, Tokyo
  - Suitengu Fujita Ophthalmo Clinic, Tokyo
  - Tamagawa Eye Clinic, Tokyo
  - Tokiwadai Muranaka Eye Clinic, Tokyo
  - Ueda Eye Clinic, Tokyo
  - Watanabe Eye Clinic, Tokyo
  - IMAI Eye Clinic, Yamanashi

IPD SHARING:
Plan to Share IPD: No